CLINICAL TRIAL: NCT04397146
Title: Palatability and Satiating Effects of Oral Nutrition Supplements as Perceived by Independently Living Older Adults
Brief Title: Palatability and Perceived Satiety of Oral Nutrition Supplements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University and Research (Other)
Collaborators: Fonterra (Europe) Cooperatie U.A. (Unknown)
Responsible Party: Principal Investigator, Diederik Esser, project leader clinical trials, Wageningen University and Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL70308.081.19
Record Dates: First submitted 2020-01-07; First posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Sensory Evaluation; Perceived Satiety

STUDY DESIGN:
Intervention Model Description: Each study participant evaluates 8 different ONS products on palatability and perceived satiety
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-blind sensory and satiety evaluation (Experimental): In total 8 different ONS products are consumed and evaluated, each product on a separate test day. The order of products is randomized between study participants.
  Interventions: Dietary Supplement: Oral Nutrition Supplement (ONS)

INTERVENTIONS:
Dietary Supplement: Oral Nutrition Supplement (ONS) — Consumption of a portion of 300-320kcal (based on a standard single serve for ONS products) with a two hour follow-up. Products include: 2 Prototype Oral Nutrition Supplements (ONS) with 2.4kcal/ml and respectively 9.6% protein and 14.4% protein; 6 Commercially available Oral Nutrition Supplements with varying energy and protein levels.

SUMMARY:
The objective of the study is to evaluate palatability (primary objective) and perceived satiating effects (secondary objective) of two Oral Nutrition Supplements (ONS) prototypes and six commercially available ONS products. The products are matched on calorie content per portion.

The study is a single-blind intervention with a within-subjects design. In total 104 apparently healthy and independently living older adults aged 65 will be recruited to participate. Participants will visit the research facilities eight times in a period of one month. On each test-day participants will consume and evaluate a single product.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or over
* Apparently healthy
* Living independently

Exclusion Criteria:

* Allergies to soy, dairy or gluten
* Following a specific diet
* BMI>30 kg/m2
* Reduced kidney function
* Suffering from Alzheimer's disease, Dementia, Parkinson's Disease, Cancer, Kidney Disease or Diabetes
* Suffering from Dysphagia
* Already using oral nutritional supplements
* Receiving any medical treatment that is known to reduce the taste or sense of smell
* Current smokers
* Participation in another clinical trial at the same time

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 104 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Liking | Immediately after consumption of one sip of the ONS product
  Questionnaire evaluating overall liking, liking of taste, liking of creaminess, liking of sweetness, liking of thickness and liking of aftertaste on a 11-points categorical scale ranging from 1='do not like at all' to 11='like very much'
Liking | Immediately after finishing consumption of a full portion of the ONS product
  Questionnaire evaluating overall liking, liking of taste, liking of thickness and liking of aftertaste on a 11-points categorical scale ranging from 1='do not like at all' to 11='like very much'

SECONDARY OUTCOMES:
Satiety | Before consumption of the ONS product
  Feelings of satiety will be evaluated using a standardized questionnaire covering hunger (3 items), thirst (2 items) and fullness (1 item). Each item is answered on a 11-points categorical scale ranging from 1='not at all' to 11='very much'
Satiety | Immediately after finishing consumption of a full portion of the ONS product
  Feelings of satiety will be evaluated using a standardized questionnaire covering hunger (3 items), thirst (2 items) and fullness (1 item). Each item is answered on a 11-points categorical scale ranging from 1='not at all' to 11='very much'
Satiety | 1 hour after finishing consumption of a full portion of the ONS product
  Feelings of satiety will be evaluated using a standardized questionnaire covering hunger (3 items), thirst (2 items) and fullness (1 item). Each item is answered on a 11-points categorical scale ranging from 1='not at all' to 11='very much'
Satiety | 2 hours after finishing consumption of a full portion of the ONS product
  Feelings of satiety will be evaluated using a standardized questionnaire covering hunger (3 items), thirst (2 items) and fullness (1 item). Each item is answered on a 11-points categorical scale ranging from 1='not at all' to 11='very much'

CONTACTS AND LOCATIONS:
Locations (1):
- Stichting Wageningen Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No